CLINICAL TRIAL: NCT04632628
Title: Web-based Cognitive Behavioral Treatment for Insomnia in Dementia Caregivers
Acronym: NiteCAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Christina McCrae, Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017125
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Insomnia Chronic; Dementia
Keywords: Dementia Caregiver; Sleep; Behavioral Interventions; Online Behavioral Intervention; Insomnia; Dementia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NiteCAPP: Online Cognitive Behavioral Therapy for Insomnia (Experimental): This is a pilot trial with one treatment condition (CBT-I).
  Interventions: Behavioral: Web-based Cognitive Behavior Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Web-based Cognitive Behavior Therapy for Insomnia (CBT-I) — Participants will complete 4 web-based CBT- I sessions. Lesson 1: Sleep Hygiene and Stimulus Control Lesson 2: Sleep Restriction and Relaxation Strategies Lesson 3: Identifying and Restructuring Dysfunction Thoughts Lesson 4: Practical Recommendations, Review, and Maintenance of Change

SUMMARY:
Over the next 30 years, more than 10 million persons living with dementia in the United States will receive care at home from an unpaid and untrained family caregiver. At home care is preferred by caregivers and persons with dementia alike, but increases the caregiver's risk of insomnia and related negative health outcomes, including depression, anxiety, cognitive disturbances and poor quality of life. Cognitive behavioral therapy for insomnia (CBT-I) is a highly effective and established evidence based treatment for adults of all ages. Although relatively understudied in dementia caregivers, the research by our group and others suggests CBT-I is also efficacious in caregivers. Our team developed a brief (4 session) CBT-I protocol specifically adapted for dementia caregivers (CBT-I) and has shown in person and remote (i.e. telehealth) delivery of this protocol significantly reduces insomnia symptoms and improves mood (moderate to large effects). Given demands on caregivers' time and limited availability of trained CBT-I providers, a web-based version of CBT-I (WebCBT-I; the online treatment will be called NiteCAPP) is needed to increase the accessibility of this efficacious treatment. WebCBT-I will allow for flexible at home scheduling, and the skills needed to monitor caregiver treatment progress can be quickly and efficiently taught to healthcare providers. The overarching goal of this project is to develop and test WebCBT-I in caregivers of persons with dementia.

Objectives

1. To examine the clinical and health characteristics, including sleep, pain, fatigue, cognitive abilities, and cardiovascular health in dementia caregivers with insomnia.
2. To examine changes in the primary clinical outcomes, including complaints of poor sleep, and fatigue.
3. To examine changes in the secondary clinical outcomes, including mood, daytime functioning, cognitive functioning, and cardiovascular health.
4. To examine the mechanistic variables, including arousal (heart rate variability, HRV).

ELIGIBILITY:
CAREGIVER

Inclusion Criteria:

* 18+ yrs
* Dementia caregiver living with person with dementia
* willing to be randomized, 4. read/understand English
* insomnia diagnosis
* no prescribed or over-the-counter sleep meds or stabilized 6+ weeks.

Insomnia:

* complaints for 6+ mos
* adequate opportunity and circumstances for sleep
* 1+ of the following: difficulty falling asleep, staying asleep, or waking too early
* daytime dysfunction (mood, cognitive, social, occupational) due to insomnia
* Screening interview indicates Insomnia Severity Index score ≥11 or Insomnia Severity Index score 9-10
* baseline diaries indicate >30 mins of sleep onset latency or wake after sleep onset on 3+ nts.

Exclusion Criteria:

* unable to consent
* cognitive impairment [Telephone Interview for Cognitive Status (TICS) <25 or Mini Mental State Examination (MMSE) <26]
* sleep disorder other than insomnia [i.e., sleep apnea (apnea/hypopnea index, AHI >15)]
* bipolar or seizure disorder
* other major psychopathology except depression or anxiety (e.g., suicidal ideation/intent, psychosis)
* severe untreated psychiatric comorbidity
* psychotropic or other medications (e.g., beta-blockers) that alter sleep
* non-pharmacological tx for sleep or mood outside current trial.

PERSONS WITH DEMENTIA

Inclusion Criteria:

* 18+ yrs
* Persons with dementia living with caregiver
* Have an eligible caregiver
* willing to be randomized

Exclusion Criteria:

• Person with dementia or legally authorized representative is unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Daily Electronic Sleep and Pain Diaries - Sleep Onset Latency | 6 weeks
  Subjective sleep onset latency (time to fall asleep)
Daily Electronic Sleep and Pain Diaries - Wake-time After Sleep Onset | 6 weeks
  Subjective time awake after sleep onset
Daily Electronic Sleep and Pain Diaries - Total Sleep Time | 6 weeks
  Subjective total sleep time
Daily Electronic Sleep and Pain Diaries - Sleep Efficiency | 6 weeks
  Subjective sleep efficiency
Daily Electronic Sleep and Pain Diaries - Pain Intensity & Unpleasantness | 6 weeks
  Pain Intensity & Unpleasantness
Daily Electronic Sleep and Pain Diaries - Medication Consumption | 6 weeks
  Sleep and pain medication consumption
Objective Daily Sleep Actiwatch-2 - Sleep Onset Latency | 6 weeks
  Objective sleep onset latency (time to fall asleep)
Objective Daily Sleep Actiwatch-2 - Wake-time After Sleep Onset | 6 weeks
  Objective time awake after sleep onset
Objective Daily Sleep Actiwatch-2 - Total Sleep Time | 6 weeks
  Objective total sleep time
Objective Daily Sleep Actiwatch-2 - Sleep Efficiency | 6 weeks
  Objective sleep efficiency
Insomnia Severity Index | 6 weeks
  Insomnia severity measurement; min: 0 max:28; higher score means greater insomnia severity

SECONDARY OUTCOMES:
State Trait Anxiety Inventory (STAI-Y1) | 6 weeks
  Assessment of anxiety symptoms - min: 0 max:60; higher score means higher anxiety
Beck Depression Inventory Second Edition (BDI- II) | 6 weeks
  Depressive symptom assessment - min: 0 max: 63; Higher score means higher severity of depression
Perceived Stress Scale (PSS) | 6 weeks
  Perception of stress - min: 0; max:40 - higher scores indicate higher perceived stress
Kingston Caregiver Stress Scale | 6 weeks
  Caregiver stress measurement - min:10 max:50 - higher score indicates higher caregiver stress
Dysfunctional Attitudes/Beliefs about Sleep (DBAS) | 6 weeks
  evaluates sleep-related beliefs, expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues - higher scores indicates more dysfunctional beliefs and attitudes
Caregiver Functional Unit Scale | 6 weeks
  Assessment of the stability of the patient-caregiver dyad - higher score indicates lower stability
Online Cognitive Assessment - Stroop | 6 weeks
  Determine level of cognitive functioning
Online Cognitive Assessment - Sternberg | 6 weeks
  Determine level of cognitive functioning
Online Cognitive Assessment - Wisconsin Card Sorting Task | 6 weeks
  Determine level of cognitive functioning
Cognitive Failures Questionnaire | 6 weeks
  Self-reported failures in perception, memory, and motor function - min:0 max: 100 - higher score indicates greater cognitive failure
Dementia Patient's Caregiver Quality of Life Scale | 6 weeks
  Assessment of caregiver quality of life - min: 0 max:100 - higher score indicates good quality of life
Zarit Burden Scale | 6 weeks
  Caregiver burden measurement - min: 0 max: 48 - higher score indicated higher caregiver burden

CONTACTS AND LOCATIONS:
Overall Officials: Christina McCrae, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

REFERENCES:
- [Background] Rowe MA, McCrae CS, Campbell JM, Benito AP, Cheng J. Sleep pattern differences between older adult dementia caregivers and older adult noncaregivers using objective and subjective measures. J Clin Sleep Med. 2008 Aug 15;4(4):362-9. PMID 18763429
- [Background] Fonareva I, Amen AM, Zajdel DP, Ellingson RM, Oken BS. Assessing sleep architecture in dementia caregivers at home using an ambulatory polysomnographic system. J Geriatr Psychiatry Neurol. 2011 Mar;24(1):50-9. doi: 10.1177/0891988710397548. PMID 21320949
- [Background] Beaudreau SA, Spira AP, Gray HL, Depp CA, Long J, Rothkopf M, Gallagher-Thompson D. The relationship between objectively measured sleep disturbance and dementia family caregiver distress and burden. J Geriatr Psychiatry Neurol. 2008 Sep;21(3):159-65. doi: 10.1177/0891988708316857. Epub 2008 May 23. PMID 18503035
- [Background] Creese J, Bedard M, Brazil K, Chambers L. Sleep disturbances in spousal caregivers of individuals with Alzheimer's disease. Int Psychogeriatr. 2008 Feb;20(1):149-61. doi: 10.1017/S1041610207005339. Epub 2007 Apr 30. PMID 17466086
- [Background] McCurry SM, Logsdon RG, Teri L, Vitiello MV. Sleep disturbances in caregivers of persons with dementia: contributing factors and treatment implications. Sleep Med Rev. 2007 Apr;11(2):143-53. doi: 10.1016/j.smrv.2006.09.002. Epub 2007 Feb 6. PMID 17287134
- [Background] McCrae CS, Wilson NM, Lichstein KL, Durrence HH, Taylor DJ, Bush AJ, Riedel BW. 'Young old' and 'old old' poor sleepers with and without insomnia complaints. J Psychosom Res. 2003 Jan;54(1):11-9. doi: 10.1016/s0022-3999(02)00543-3. PMID 12505551
- [Background] Mahoney DF. Vigilance. Evolution and definition for caregivers of family members with Alzheimer's disease. J Gerontol Nurs. 2003 Aug;29(8):24-30. doi: 10.3928/0098-9134-20030801-07. PMID 13677157
- [Background] McCrae CS, Curtis AF, Williams JM, Dautovich ND, McNamara JPH, Stripling A, Dzierzewski JM, Chan WS, Berry RB, McCoy KJM, Marsiske M. Efficacy of brief behavioral treatment for insomnia in older adults: examination of sleep, mood, and cognitive outcomes. Sleep Med. 2018 Nov;51:153-166. doi: 10.1016/j.sleep.2018.05.018. Epub 2018 Jun 2. PMID 30195661
- [Background] Edinger JD, Wohlgemuth WK, Krystal AD, Rice JR. Behavioral insomnia therapy for fibromyalgia patients: a randomized clinical trial. Arch Intern Med. 2005 Nov 28;165(21):2527-35. doi: 10.1001/archinte.165.21.2527. PMID 16314551
- [Background] McCrae CS, McGovern R, Lukefahr R, Stripling AM. Research Evaluating Brief Behavioral Sleep Treatments for Rural Elderly (RESTORE): a preliminary examination of effectiveness. Am J Geriatr Psychiatry. 2007 Nov;15(11):979-82. doi: 10.1097/JGP.0b013e31813547e6. PMID 17974868
- [Background] Glass J, Lanctot KL, Herrmann N, Sproule BA, Busto UE. Sedative hypnotics in older people with insomnia: meta-analysis of risks and benefits. BMJ. 2005 Nov 19;331(7526):1169. doi: 10.1136/bmj.38623.768588.47. Epub 2005 Nov 11. PMID 16284208
- [Background] Allain H, Bentue-Ferrer D, Polard E, Akwa Y, Patat A. Postural instability and consequent falls and hip fractures associated with use of hypnotics in the elderly: a comparative review. Drugs Aging. 2005;22(9):749-65. doi: 10.2165/00002512-200522090-00004. PMID 16156679
- [Background] Trauer JM, Qian MY, Doyle JS, Rajaratnam SM, Cunnington D. Cognitive Behavioral Therapy for Chronic Insomnia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Aug 4;163(3):191-204. doi: 10.7326/M14-2841. PMID 26054060
- [Background] Bertisch SM, Herzig SJ, Winkelman JW, Buettner C. National use of prescription medications for insomnia: NHANES 1999-2010. Sleep. 2014 Feb 1;37(2):343-9. doi: 10.5665/sleep.3410. PMID 24497662
- [Background] Qaseem A, Kansagara D, Forciea MA, Cooke M, Denberg TD; Clinical Guidelines Committee of the American College of Physicians. Management of Chronic Insomnia Disorder in Adults: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2016 Jul 19;165(2):125-33. doi: 10.7326/M15-2175. Epub 2016 May 3. PMID 27136449
- [Background] McCurry SM, Gibbons LE, Logsdon RG, Vitiello MV, Teri L. Insomnia In Caregivers Of Persons With Dementia: Who Is At Risk And What Can Be Done About It? Sleep Med Clin. 2009 Dec 1;4(4):519-526. doi: 10.1016/j.jsmc.2009.07.005. PMID 20046806
- [Background] McCrae CS, Tierney CG, McNamara JP. Behavioral intervention for insomnia: Future directions for nontraditional caregivers at various stages of care. Clinical gerontologist. 2006;29(2):95-114.
- [Background] McCurry SM, Logsdon RG, Vitiello MV, Teri L. Successful behavioral treatment for reported sleep problems in elderly caregivers of dementia patients: a controlled study. J Gerontol B Psychol Sci Soc Sci. 1998 Mar;53(2):P122-9. doi: 10.1093/geronb/53b.2.p122. PMID 9520929
- [Background] McCrae CS, Tierney CG, McNamara JP. Behavioral Intervention for Insomnia: Future Directions for Nontraditional Caregivers at Various Stages of Care. Clinical Geropsychologist. 2005;29(2):95-115.
- [Background] Lichstein KL, Wilson NM, Johnson CT. Psychological treatment of secondary insomnia. Psychol Aging. 2000 Jun;15(2):232-40. doi: 10.1037//0882-7974.15.2.232. PMID 10879578
- [Background] Grant JS, Bartolucci AA, Elliot TR, Giger JN. Sociodemographic, physical, and psychosocial characteristics of depressed and non-depressed family caregivers of stroke survivors. Brain Inj. 2000 Dec;14(12):1089-100. doi: 10.1080/02699050050203586. PMID 11147581
- [Background] Nezu AM, Nezu CM, Perri MG. Psychotherapy for adults within a problem-solving framework: Focus on depression. J Cogn Psychother. 1990;4(3):247-256.
- [Background] Pinquart M, Sorensen S. Differences between caregivers and noncaregivers in psychological health and physical health: a meta-analysis. Psychol Aging. 2003 Jun;18(2):250-67. doi: 10.1037/0882-7974.18.2.250. PMID 12825775
- [Background] Schulz R, Martire LM. Family caregiving of persons with dementia: prevalence, health effects, and support strategies. Am J Geriatr Psychiatry. 2004 May-Jun;12(3):240-9. PMID 15126224
- [Background] Sakurai S, Onishi J, Hirai M. Impaired autonomic nervous system activity during sleep in family caregivers of ambulatory dementia patients in Japan. Biol Res Nurs. 2015 Jan;17(1):21-8. doi: 10.1177/1099800414524050. Epub 2014 Feb 25. PMID 25504947
- [Background] Hasuo H, Kanbara K, Sakuma H, Yoshida K, Uchitani K, Fukunaga M. Self-Care System for Family Caregivers of Cancer Patients Using Resonant Breathing with a Portable Home Device: A Randomized Open-Label Study. J Palliat Med. 2019 Jan;22(1):18-24. doi: 10.1089/jpm.2018.0230. Epub 2018 Sep 5. PMID 30183463
- [Background] Lee KC, Yiin JJ, Chao YF. Effect of integrated caregiver support on caregiver burden for people taking care of people with cancer at the end of life: A cohort and quasi-experimental clinical trial. Int J Nurs Stud. 2016 Apr;56:17-26. doi: 10.1016/j.ijnurstu.2016.01.002. Epub 2016 Jan 12. PMID 26794928
- [Background] Schulz R, O'Brien AT, Bookwala J, Fleissner K. Psychiatric and physical morbidity effects of dementia caregiving: prevalence, correlates, and causes. Gerontologist. 1995 Dec;35(6):771-91. doi: 10.1093/geront/35.6.771. PMID 8557205
- [Background] Yates ME, Tennstedt S, Chang BH. Contributors to and mediators of psychological well-being for informal caregivers. J Gerontol B Psychol Sci Soc Sci. 1999 Jan;54(1):P12-22. doi: 10.1093/geronb/54b.1.p12. PMID 9934391
- [Background] McCrae CS, Dzierzewski JM, McNamara JP, Vatthauer KE, Roth AJ, Rowe MA. Changes in Sleep Predict Changes in Affect in Older Caregivers of Individuals with Alzheimer's Dementia: A Multilevel Model Approach. J Gerontol B Psychol Sci Soc Sci. 2016 May;71(3):458-62. doi: 10.1093/geronb/gbu162. Epub 2014 Nov 26. PMID 25429026
- [Background] Caswell LW, Vitaliano PP, Croyle KL, Scanlan JM, Zhang J, Daruwala A. Negative associations of chronic stress and cognitive performance in older adult spouse caregivers. Exp Aging Res. 2003 Jul-Sep;29(3):303-18. doi: 10.1080/03610730303721. PMID 12775440
- [Background] Vitaliano PP, Zhang J, Young HM, Caswell LW, Scanlan JM, Echeverria D. Depressed mood mediates decline in cognitive processing speed in caregivers. Gerontologist. 2009 Feb;49(1):12-22. doi: 10.1093/geront/gnp004. Epub 2009 Mar 18. PMID 19363000
- [Background] Mackenzie CS, Smith MC, Hasher L, Leach L, Behl P. Cognitive functioning under stress: evidence from informal caregivers of palliative patients. J Palliat Med. 2007 Jun;10(3):749-58. doi: 10.1089/jpm.2006.0171. PMID 17592987
- [Background] Oken BS, Fonareva I, Wahbeh H. Stress-related cognitive dysfunction in dementia caregivers. J Geriatr Psychiatry Neurol. 2011 Dec;24(4):191-8. doi: 10.1177/0891988711422524. PMID 22228825
- [Background] Astell A, Alm N, Gowans G, Ellis M, Dye R, Vaughan P. Involving older people with dementia and their carers in designing computer based support systems: some methodological considerations. Universal Access in the Information Society. 2009;8(1):49.
- [Background] Lichstein KL, Riedel BW, Grieve R. Fair tests of clinical trials: A treatment implementation model. Advances in Behaviour Research and Therapy. 1994;16(1):1-29.
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hopkins R, Kilik L. Kingston Caregiver Stress Scale administration and interpretation manual. Kingston, Canada: Geriatric Psychiatry Programme, Providence Care, Mental...; 2012.
- [Background] Morin CM. Insomnia: Psychological assessment and management.Guilford Press; 1993.
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Slotkin J, Kallen M, Griffith J, et al. NIH toolbox technical manual. Bethesda, MD: National Institutes of Health. 2012.
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Thomas P, Lalloue F, Preux PM, Hazif-Thomas C, Pariel S, Inscale R, Belmin J, Clement JP. Dementia patients caregivers quality of life: the PIXEL study. Int J Geriatr Psychiatry. 2006 Jan;21(1):50-6. doi: 10.1002/gps.1422. PMID 16323256
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Beck AT, Steer RA, Garbin MG. Beck Depression Inventory-Second Edition.San Antonio, TX: The Psychological Corporation; 1996.
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA. State-Trait Anxiety Inventory, Form Y.Palo Alto, CA: Consulting Psychologists Press; 1983.
- [Derived] McCrae CS, Curtis AF, Stearns MA, Nair N, Golzy M, Shenker JI, Beversdorf DQ, Cottle A, Rowe MA. Development and Initial Evaluation of Web-Based Cognitive Behavioral Therapy for Insomnia in Rural Family Caregivers of People With Dementia (NiteCAPP): Mixed Methods Study. JMIR Aging. 2023 Aug 24;6:e45859. doi: 10.2196/45859. PMID 37616032